CLINICAL TRIAL: NCT02980744
Title: The Feasibility of a Home-based Transition Intervention to Reduce Sedentary Behaviour and Improve Function Within the First Six Months After Stroke: STand Up Frequently From Stroke Trial
Brief Title: A Home-based Intervention to Reduce Sedentary Behaviour and Improve Function After Stroke
Acronym: STUFFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Glenrose Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00053129
Record Dates: First submitted 2016-11-25; First posted 2016-12-02 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Stroke
Keywords: Stroke; Sedentary behaviour; Intervention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- STUFFS (Experimental): Participants will undergo a sedentary behaviour intervention which includes breaking up prolonged sitting by standing and walking around for 5 minutes every half-hour, standing and walking during television commercial breaks, doing 2 sets of 10 sit-to-stand transitions three times per day, and going to the kitchen to grab some drink every hour. A wrist-worn Misfit activity monitor - a motivational tool that will track adherence to the intervention will be used throughout the intervention period (i.e. 8 weeks). This device which is commercially available provides activity feedback for the user in real time.
  Interventions: Behavioral: Sedentary behaviour intervention

INTERVENTIONS:
Behavioral: Sedentary behaviour intervention — The intervention is based on socio-cognitive theory and focuses on building and increasing confidence (self-efficacy) to make a behaviour change. Output from the activity monitor (i.e. activPAL) will provide visual feedback of usual activity. Action plans targeting areas of high sedentary behaviour will be developed. A wrist-worn Misfit activity monitor is used as a self-monitoring tool throughout the intervention. This commercially available device provides activity information in real time, and sets daily targets for physical activity. A checklist will be used to address: 1) use of walking aids; 2) incidence of falls; 3) review and progression of home exercise program; and 4) quality of walking. The intervention visits will be conducted by a physical therapist.

SUMMARY:
The traditional approach to physical activity promotion in people with stroke has always emphasized activities of a moderate-to-vigorous intensity (i.e. moving enough to breathe fast and break a sweat). For many people with stroke who often have difficulty with walking, achieving that intensity of activity is difficult. The result is that people with stroke spend over 80% of their day in sedentary behaviours (too much sitting). A growing body of research shows that too much sitting has negative effects on health including larger waist circumference, unhealthy levels of blood glucose and insulin, heart disease, lower levels of functioning, and premature death.

This project tests a new approach to activity promotion that focuses on increasing light-intensity activity throughout the whole day while reducing sitting time. The new intervention is titled "STand Up Frequently From Stroke (STUFFS)" and is aimed at increasing self-confidence among people with stroke to sit less, stand up and walk around at frequent intervals during the day. Studies in the general population have shown that standing up and walking around frequently are beneficially associated with health indicators (lower waist circumference, lower blood fat and glucose levels). Encouraging people with stroke to reduce sitting and increase light-intensity activities appears feasible and sustainable and might be a first step to increase their daily energy expenditure.

DETAILED DESCRIPTION:
Background: Stroke is a leading cause of adult disability among Canadians, with about 405,000 individuals living with the effects of stroke and this number is expected to rise by 80% in the next 20 years [1]. Guidelines on activity promotion in people with stroke emphasize the attainment of 150 minutes of moderate-to-vigorous intensity activity per week [2].

Moving fast enough to 'break a sweat' is challenging for people with stroke who often have mobility deficits. Stroke survivors spend over 80% of their day in sedentary behaviours (too much sitting) [3-5]. Accumulating evidence indicates that sedentary behaviour has deleterious effects on health, regardless of exercise levels [6]. Targeting sedentary behaviour might be a feasible and sustainable way to change activity behaviour in people with stroke.

Purpose: This research aims to test the feasibility of a social cognitive theory-based intervention to reduce sedentary behaviour and improve light-intensity activity (such as standing and walking around frequently). The focus is on improving activity behaviour and will allow a systematic and staged reduction of contact with organised hospital care.

Methodological approach: Thirty-five persons with stroke will be enrolled. Outcomes including sedentary behaviour, physical activity and function will be measured at baseline (week 0), post-intervention (week 9) and follow-up (week 16). Activity behaviour (i.e. time sedentary, standing, and stepping) will be recorded for 7 days at each time point using activPAL activity monitor, validated in people with stroke [7]. Impairment from stroke will be assessed using Chedoke McMaster Stroke Assessment, which is a valid and reliable tool to measure impairment after stroke [8]. Cognitive status will be assessed using Montreal Cognitive Assessment scale, validated in stroke [9].

At the end of the intervention, feasibility outcomes such as reach (number enrolled / number eligible), retention (% enrolled who complete study), and satisfaction (exit interviews) with the program will be determined. Changes in sedentary, physical activity and functional outcomes across time (weeks 0, 9 and 16) will be tested.

Intervention: For the intervention, output from baseline activity monitoring (using activPAL activity monitor) will provide data on usual activity behaviour. Action plans targeting areas of high sedentary behaviour throughout the day will be developed. A wrist-worn activity Misfit monitor - a motivational tool that will track adherence to the intervention will be used throughout the intervention period (i.e. 8 weeks). This device provides activity feedback for the user in real time. A checklist will be used to address: 1) use of walking aids; 2) incidence of falls; 3) review and progression of home exercise program; and 4) quality of walking.

Analysis: Descriptive statistics will be used to summarize baseline data. Feasibility measurements (reach, retention, and satisfaction) will be evaluated as percentages. Changes in activity and functional outcomes across time (weeks 0, 9 and 16) will be tested using repeated measures analysis of variance (ANOVA). All analysis will be done with STATA and significance level set at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* ischemic or hemorrhagic stroke
* within 1 month of discharge from hospital
* able to stand up from a chair with or without gait aid and walk at least 5 metres
* able to understand 2-step commands

Exclusion Criteria:

* Have other neurological problems besides stroke or medically unstable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Reach | Follow-up (week 16)
  Number enrolled divided by number eligible
Retention | Follow-up (week 16)
  Percentage of those enrolled who completed the program
Satisfaction with program | Post-intervention (week 9)
  Post-intervention interviews will be conducted to assess satisfaction with the program, participants' satisfaction as a percentage will be determined.

SECONDARY OUTCOMES:
Change in sedentary time | baseline - week 0 (within one month of discharge from inpatient rehab), week 9 (post-intervention), week 16 (follow-up)
  To assess change in accelerometer-derived sedentary time from baseline to post-intervention and follow-up periods
Change in standing time | baseline - week 0 (within one month of discharge from inpatient rehab), week 9 (post-intervention), week 16 (follow-up)
  To assess change in accelerometer-derived standing time from baseline to post-intervention and follow-up periods
Change in stepping time | baseline - week 0 (within one month of discharge from inpatient rehab), week 9 (post-intervention), week 16 (follow-up)
  To assess change in accelerometer-derived stepping time from baseline to post-intervention and follow-up periods
Change in number of sit-to-stand transitions | baseline - week 0 (within one month of discharge from inpatient rehab), week 9 (post-intervention), week 16 (follow-up)
  To assess change in accelerometer-derived number of sit-to-stand transitions from baseline to post-intervention and follow-up periods
Change in resting blood pressure | baseline - week 0 (within one month of discharge from inpatient rehab), week 9 (post-intervention), week 16 (follow-up)
  To assess change in systolic and diastolic blood pressure from baseline to post-intervention and follow-up periods
Change in waist circumference | baseline - week 0 (within one month of discharge from inpatient rehab), week 9 (post-intervention), week 16 (follow-up)
  To assess change in waist circumference from baseline to post-intervention and follow-up periods
Change in gait speed | baseline - week 0 (within one month of discharge from inpatient rehab), week 9 (post-intervention), week 16 (follow-up)
  To assess change in walking speed from baseline to post-intervention and follow-up periods
Change in self-efficacy scale | baseline - week 0 (within one month of discharge from inpatient rehab), week 9 (post-intervention), week 16 (follow-up)
  To assess change in self-efficacy using Multidimensional Self-Efficacy Scale (MSES) over time from baseline to post-intervention and follow-up periods
Change in Quality-of-Life scale | baseline - week 0 (within one month of discharge from inpatient rehab), week 9 (post-intervention), week 16 (follow-up)
  To assess change in quality of life using Stroke Impact Scale from baseline to post-intervention and follow-up
Change in lower extremity impairment | baseline - week 0 (within one month of discharge from inpatient rehab), week 9 (post-intervention), week 16 (follow-up)
  To assess change in lower extremity impairment using Chedoke McMaster Stroke Assessment for leg and foot over time from baseline to post-intervention and follow-up periods
Change in cognitive scale | baseline - week 0 (within one month of discharge from inpatient rehab), week 9 (post-intervention), week 16 (follow-up)
  To assess change in cognition using Montreal Cognitive Assessment scale from baseline to post-intervention and follow-up periods

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Manns, PT, PhD, Principal Investigator — University of Alberta; Victor Ezeugwu, PT, MSc, Study Director — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data related to activPAL sedentary and activity monitoring might be shared with supervisors and other researchers

REFERENCES:
- [Background] Krueger H, Koot J, Hall RE, O'Callaghan C, Bayley M, Corbett D. Prevalence of Individuals Experiencing the Effects of Stroke in Canada: Trends and Projections. Stroke. 2015 Aug;46(8):2226-31. doi: 10.1161/STROKEAHA.115.009616. PMID 26205371
- [Background] Coutts SB, Wein TH, Lindsay MP, Buck B, Cote R, Ellis P, Foley N, Hill MD, Jaspers S, Jin AY, Kwiatkowski B, MacPhail C, McNamara-Morse D, McMurtry MS, Mysak T, Pipe A, Silver K, Smith EE, Gubitz G; Heart, and Stroke Foundation Canada Canadian Stroke Best Practices Advisory Committee. Canadian Stroke Best Practice Recommendations: secondary prevention of stroke guidelines, update 2014. Int J Stroke. 2015 Apr;10(3):282-91. doi: 10.1111/ijs.12439. Epub 2014 Dec 23. PMID 25535808
- [Background] Tieges Z, Mead G, Allerhand M, Duncan F, van Wijck F, Fitzsimons C, Greig C, Chastin S. Sedentary behavior in the first year after stroke: a longitudinal cohort study with objective measures. Arch Phys Med Rehabil. 2015 Jan;96(1):15-23. doi: 10.1016/j.apmr.2014.08.015. Epub 2014 Sep 16. PMID 25220942
- [Background] Rand D, Eng JJ, Tang PF, Jeng JS, Hung C. How active are people with stroke?: use of accelerometers to assess physical activity. Stroke. 2009 Jan;40(1):163-8. doi: 10.1161/STROKEAHA.108.523621. Epub 2008 Oct 23. PMID 18948606
- [Background] Paul L, Brewster S, Wyke S, Gill JM, Alexander G, Dybus A, Rafferty D. Physical activity profiles and sedentary behaviour in people following stroke: a cross-sectional study. Disabil Rehabil. 2016;38(4):362-7. doi: 10.3109/09638288.2015.1041615. Epub 2015 May 4. PMID 25936730
- [Background] Biswas A, Oh PI, Faulkner GE, Bajaj RR, Silver MA, Mitchell MS, Alter DA. Sedentary time and its association with risk for disease incidence, mortality, and hospitalization in adults: a systematic review and meta-analysis. Ann Intern Med. 2015 Jan 20;162(2):123-32. doi: 10.7326/M14-1651. PMID 25599350
- [Background] Taraldsen K, Askim T, Sletvold O, Einarsen EK, Bjastad KG, Indredavik B, Helbostad JL. Evaluation of a body-worn sensor system to measure physical activity in older people with impaired function. Phys Ther. 2011 Feb;91(2):277-85. doi: 10.2522/ptj.20100159. Epub 2011 Jan 6. PMID 21212377
- [Background] Gowland C, Stratford P, Ward M, Moreland J, Torresin W, Van Hullenaar S, Sanford J, Barreca S, Vanspall B, Plews N. Measuring physical impairment and disability with the Chedoke-McMaster Stroke Assessment. Stroke. 1993 Jan;24(1):58-63. doi: 10.1161/01.str.24.1.58. PMID 8418551
- [Background] Xu Q, Cao WW, Mi JH, Yu L, Lin Y, Li YS. Brief screening for mild cognitive impairment in subcortical ischemic vascular disease: a comparison study of the Montreal Cognitive Assessment with the Mini-Mental State Examination. Eur Neurol. 2014;71(3-4):106-14. doi: 10.1159/000353988. Epub 2013 Dec 10. PMID 24335198
- [Derived] Ezeugwu VE, Manns PJ. Using Intervention Mapping to develop and implement a home-based sedentary behavior change intervention after stroke. Transl Behav Med. 2020 Feb 3;10(1):87-95. doi: 10.1093/tbm/iby128. PMID 30566661
- [Derived] Ezeugwu VE, Manns PJ. The Feasibility and Longitudinal Effects of a Home-Based Sedentary Behavior Change Intervention After Stroke. Arch Phys Med Rehabil. 2018 Dec;99(12):2540-2547. doi: 10.1016/j.apmr.2018.06.014. Epub 2018 Jul 5. PMID 29981314